CLINICAL TRIAL: NCT04725292
Title: Pseudoepitheliomatous Hyperplasia of the Penis a Very Rare Disease in Egypt
Brief Title: Rare Benign Lesion of Peins
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, chief resident of urology, Assiut University
Other Study IDs: penis skin lesion
Record Dates: First submitted 2021-01-16; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Skin Diseases; Penile Diseases
MeSH Terms: conditions — Skin Diseases; Penile Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PEKMB was first named and described by Lortat-Jacob & Civatte in 1961 and by Bart & Kopf later. This rare condition is mostly reported in elderly males. The keratotic scales is usually micaceous and resembles psoriasis. Most patients are above 50 years of age and are circumcised later in life, but also reported in younger age group. This mica like scales contains keratin which gets dissolved in 10% potassium hydroxide solution. Disease progression may lead to phimosis. Differential diagnosis of this disease entity include moniliasis, wart, psoriasis ,penile horn, circinate balanitis, erythroplasia of Queyrat, squamous cell epithelioma and verrucous carcinoma. It is primarily a benign entity, it is capable of invasiveness. Bart and Kopf considered it to be in intermediate stage between benign hyperplasia and squamous cell carcinoma. However, the histological spectrum can range from hypertrophic-hyperplastic penile dystrophy to verrucous carcinoma. Fibro sarcoma has been reported developing in a same patient. Etiology is unclear. Despite search for a viral agent, Human Papilloma Virus (HPV) has not been demonstrated and its role in pathogenesis or its transformation to verrucous carcinoma has been proved. The treatment of PEKMB should be conservative when there is no histological evidence of malignancy. All such patients should be followed up. Treatment choices include potent topical steroids, topical 5% 5-flurouracil cream1, 2, cryotherapy, radiotherapy and shaving biopsy plus electro coagulation. When frank malignancy is observed, excision with wide margin is the rule.

ELIGIBILITY:
Inclusion Criteria:

* 40 years
* failed medical treatment

Exclusion Criteria:

* psoriasis
* allergy
* trauma

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — case report
Study Population: male healthy married
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
improvement of the skin lesion | 1 month after treatment
  drugs will be given to patient then the effect ,either improvement or worsening will be noticied
improvement of associated lesion | 1 month after drug given
  patient complained of difficulty and burning micturition which will be seen after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit Medical School, Asyut, Assuit, Egypt